CLINICAL TRIAL: NCT04600154
Title: Effects of MS-20 on Gut Microbiota and Risk/Severity of Cachexia in Patients Receiving Chemotherapy for Pancreatic Cancer
Brief Title: MS-20 on Gut Microbiota and Risk/Severity of Cachexia in Pancreatic Cancer Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Collaborators: Microbio Co Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 202004004MIPC
Record Dates: First submitted 2020-09-21; First posted 2020-10-23 (Actual); Last update posted 2023-01-19 (Actual); Status verified 2023-01

CONDITIONS: Pancreatic Cancer; Cachexia; Chemotherapy Effect
Keywords: Pancreatic cancer; Cachexia; Randomized controlled trial; Microbiota
MeSH Terms: conditions — Pancreatic Neoplasms; Cachexia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MS-20 (Experimental): 4ml, twice, daily
  Interventions: Drug: MS-20
- Placebo (Placebo Comparator): 4ml, twice, daily
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: MS-20 — Specific fraction from fermented soy milk
  Other Names: Chemo young oral solution
  Arms: MS-20
Other: Placebo — Fermented soy milk without active component
  Arms: Placebo

SUMMARY:
Cachexia has been recognized as a direct cause of reduced quality of life complicating in cancer patients. Patients with pancreatic cancer have the highest prevalence in developing severe degrees of cachexia. Providing supportive therapies for these patients may provide a lot of benefit on overarching quality of life and improve overall survival.

MS-20 is indicated for treating the symptom of fatigue and loss of appetite induced by chemotherapy in cancer patients. According to the result from pre-clinical study, MS-20 may have potential to attenuate or suppress the resistant phenomena of chemotherapy via alternating gut microbiota profile.

In this study, MS-20 effects on on gut microbiota and risk/severity of cachexia will be analyzed in pancreatic cancer patients who under combination therapy with chemotherapy and MS-20.

DETAILED DESCRIPTION:
This is a double-blind, placebo-controlled, investigator-initiated randomized trial to evaluate the effects of MS-20 on gut microbiota and risk/severity of cachexia in patients receiving chemotherapy for pancreatic cancer. Approximately 40 subjects who meet the criteria will be enrolled into the study. The total of study comprises of a 28 days screening period, a 12-week treatment period and a 8-week follow-up period.

Potential candidates should provide signed informed consent forms before starting any screening activities. MS-20 or placebo will be orally administered twice per day in treatment period. All medications (especially antibiotics) should be recorded and documented during the study period.

The investigator may withdraw a subject from the study if any of the following conditions occurs:

1. Subjects who experiences a serious adverse event (SAE) or intolerable adverse event (AE), or laboratory safety assessments reveal clinically significant hematological or biochemical changes from baseline values.
2. The subject would like to withdraw consent and discontinue from the study at any time, for any reason, without any influence on further treatment. (Patients who withdraw or terminate early from study should proceed to EOT visit for safety evaluation.)

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects aged between 20 and 75 years old.
2. Patients with histologically- or cytologically-confirmed unresectable locally advanced or metastatic pancreatic ductal adenocarcinoma (PDAC) who plan to receive gemcitabine alone or in combination with other chemotherapeutic agents.
3. ECOG (Eastern Cooperative Oncology Group Performance status) scale between 0 and 2.
4. Female subjects of childbearing potential must use at least two forms of birth control. Subjects who are postmenopausal (defined as amenorrhea for 12 consecutive months) , surgically sterilized (ie, hysterectomy, bilateral oophorectomy, or bilateral tubal ligation), or have abnormalities of the reproductive tract will be considered as having no childbearing potential.
5. The subject is able to provide written informed consent by himself/herself and agrees to comply with all protocol requirements.
6. The subject agrees to comply with the following two requirements:

   1. comply with all follow-up visit requirements according to the trial protocol.
   2. comply with all requirement regarding fecal samples collection, storage and delivery according to the trial protocol.

Exclusion Criteria:

1. The subject has soybean allergy.
2. The subject is pregnant or lactating.
3. The subject has received or is receiving chemotherapy.
4. The subject has received any antibiotic, antifungals or antivirals (excluding topical agents and antiviral prophylaxis for hepatitis B virus) within 14 days prior to visit 2 (Day 1).
5. The subject has a clinically significant, currently active or underlying diarrhea (soft or loose stools more than three times in 24 hours) of infectious etiologies.
6. The subject has received any steroids, immunosuppressant or anti-inflammation drugs within 14 days prior to visit 2 (Day 1)..
7. The subject has received probiotics or prebiotics within 14 days prior to visit 2 (Day 1).
8. The subject has abnormal organ and bone marrow function as defined below:

   1. Patients with abnormal liver function tests (serum bilirubin level ≧ 2 times upper limit of normal (ULN), aspartate transaminase (AST) or alanine transaminase (ALT) ≧ 3.0 X ULN).
   2. Patients with renal disease or renal dysfunction (serum creatinine ≧ 1.5 X ULN) or estimated glomerular filtration rate (eGFR)< 50 mL/min/1.73 m2.
9. The subject has active inflammatory bowel disease or gastric ulcer.
10. The subject currently is participating in studies involving other investigational drugs, medical devices, functional foods, or cosmetics.
11. The subject is considered by the investigator as not suitable for the trial.
12. The subject is judged by the investigator as not suitable for the trial due to concerns about possible non-compliance or severe concomitant illnesses.

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2021-08-10 (Actual); Primary Completion 2023-06-30 (Estimated); Study Completion 2023-06-30 (Estimated)

PRIMARY OUTCOMES:
Change in cachexia staging score from baseline | baseline to 12th week
  Cachexia staging score: a score to gauge the severity of cachexia: non-cachexia (0-2), pre-cachexia (3-4), cachexia (5-8), and refractory cachexia (9-12)

SECONDARY OUTCOMES:
Change in lumbar skeletal muscle index from baseline | baseline to 12th week
  Lumbar skeletal muscle index (SMI) is calculated as the mean of sum of cross-sectional areas of skeletal muscles on two consecutive CT images containing the third lumbar vertebra
QLQ-C30 Global health status/QoL | 12th week
  Linear transformation of Global health status/QoL score of QLQ-C30

OTHER OUTCOMES:
Progression free survival | From enrollment to progressive disease, or censored at end of study (20th week)
  Time from enrollment to progressive disease (PD) as assessed by Response Evaluation Criteria In Solid Tumours (RECIST) 1.1

CONTACTS AND LOCATIONS:
Overall Officials: Wei-Chih Liao, MD/PhD, Principal Investigator — Department of Internal Medicine, National Taiwan University Hospital
Locations (1):
- Department of Internal Medicine, National Taiwan University Hospital, Taipei, Taiwan